CLINICAL TRIAL: NCT06091865
Title: A Phase 3, Open Label, Randomized Study Comparing the Efficacy and Safety of Odronextamab (REGN1979), an Anti-CD20 × Anti-CD3 Bispecific Antibody, in Combination With CHOP (ODRO-CHOP) Versus Rituximab in Combination With CHOP (R-CHOP) in Previously Untreated Participants With Diffuse Large B-cell Lymphoma (DLBCL) (OLYMPIA-3)
Brief Title: A Study to Compare How Well Odronextamab Combined With Chemotherapy Works and How Safe it is Against Rituximab Combined With Chemotherapy, in Adult Patients With Previously Untreated Diffuse Large B-cell Lymphoma
Acronym: OLYMPIA-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R1979-ONC-2105; 2022-502785-25-00 (EU CTIS Number)
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Large B-cell Lymphoma (DLBCL)
Keywords: Non-Hodgkin Lymphomas (NHL); B-cell Non-Hodgkin Lymphomas (B-NHL); Diffuse Large B-cell Lymphoma; Odronextamab; Anti-CD20 × anti-CD3 bispecific antibody
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Odronextamab + CHOP (Experimental): Part 1, includes dose escalation (Part 1A), and randomized exploration of 2 regimens of odronextamab -cyclophosphamide, doxorubicin, vincristine, prednisone (Odro-CHOP) dose optimization (Part 1B).
  Interventions: Drug: Odronextamab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone/Prednisolone
- Rituximab + CHOP (Active Comparator): Part 2 is the randomized controlled portion, participants will receive either Odro-CHOP or R-CHOP.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone/Prednisolone

INTERVENTIONS:
Drug: Odronextamab — Odronextamab will be administered by intravenous (IV) infusion
  Other Names: REGN1979; Ordspono™
  Arms: Odronextamab + CHOP
Drug: Rituximab — Rituximab will be administered IV, or subcutaneously (SC)
  Other Names: RITUXAN®
  Arms: Rituximab + CHOP
Drug: Cyclophosphamide — Cyclophosphamide will be administered IV as part of chemotherapy
  Other Names: Cytoxan®
Drug: Doxorubicin — Doxorubicin will be administered IV as part of chemotherapy
  Other Names: Adriamycin®
Drug: Vincristine — Vincristine will be administered IV as part of chemotherapy
  Other Names: Oncovin®; Vincasar PFS®
Drug: Prednisone/Prednisolone — Prednisone or prednisolone will be administered orally (PO) as part of chemotherapy
  Other Names: Deltasone®/OMNIPRED®

SUMMARY:
This study is researching an experimental drug called odronextamab, referred to as study drug, when used in combination with chemotherapy. The study is focused on patients with Diffuse Large B-cell Lymphoma (DLBCL) that have not been treated before (called "previously untreated"). Patients with DLBCL that have come back after treatment (called "relapsed"), or have not responded to treatment (called "refractory"), can also participate in this study.

This study will be made up of Part 1A, Part 1B, and Part 2.The aim of Part 1A and Part 1B of the study is to see how safe and tolerable the study drug in combination with chemotherapy is and to determine the dose and schedule of the study drug to be combined with chemotherapy in Part 2 of the study.

The aim of Part 2 of the study is to see how effective the combination of the study drug with chemotherapy is in comparison with the combination of rituximab (the comparator drug), and chemotherapy, the current standard of care treatment approved for DLBCL. Standard of care means the usual medication expected and used when receiving treatment for a condition.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug when combined with chemotherapy
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the study drug less effective or could lead to side effects)
* The impact from the study drug on quality of life and ability to complete routine daily activities

ELIGIBILITY:
Key Inclusion Criteria:

1. Previously untreated participants for lymphoma with documented Cluster of Differentiation 20+ (CD20+) DLBCL, as described in the protocol OR relapsed or refractory DLBCL, for whom next available standard of care therapy is not available or deemed ineligible according to the investigator (Part 1A only)
2. Measurable disease with at least one nodal lesion or at least one extranodal lesion, as described in the protocol
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤2
4. Life expectancy ≥ 12 months
5. International Prognostic Index (IPI) of 3 to 5 (part 1 only) and ≥2 (part 2) for untreated DLBCL only
6. Adequate hematologic and organ function, as defined in the protocol.

Key Exclusion Criteria:

1. Primary Central Nervous System (CNS) lymphoma or known involvement by non-primary CNS NHL and history or current relevant CNS pathology
2. Another active malignancy, significant active disease or medical condition, as described in the protocol
3. Peripheral neuropathy Grade ≥3
4. Treatment with any systemic anti-lymphoma therapy, except for participants with Relapsed/Refractory (R/R) DLBCL and participants with DLBCL transformed from an indolent lymphoma after treatment with systemic anti-lymphoma therapy.
5. Any other therapy or investigational treatment within 28 days or 5 half-lives of the drug, whichever is shorter, prior to the start of study treatment
6. Recent major surgery, prior organ transplantation, or standard radiotherapy, as described in the protocol
7. Allergy/hypersensitivity to study drugs, as described in the protocol
8. Infections such as any active infection (bacterial, viral, fungal, mycobacterial, parasitic or other), active Coronavirus Disease (COVID-19) infection, uncontrolled infection with Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV), Cytomegalovirus (CMV) infection, as described in the protocol.

Note: Other protocol-defined Inclusion/ Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 904 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2029-09-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | Up to 35 days
  Part 1A
Incidence of Treatment Emergent Adverse Events (TEAEs) | Up to 2 years
  Part 1
Severity of TEAEs | Up to 2 years
  Part 1
Progression Free Survival (PFS), assessed by Independent Central Review (ICR) | Up to 5 years
  Part 2

SECONDARY OUTCOMES:
Event-Free Survival (EFS) assessed by ICR | Up to 5 years
  Part 2
Complete Response (CR) assessed by ICR | Up to 22 weeks
  Part 2
Overall Survival (OS) | Up to 5 years
  Part 2
Best Overall Response (BOR) as assessed by local investigators | Up to 22 weeks
  Part 1 and Part 2
CR as assessed by local investigators | Up to 22 weeks
  Part 1 and Part 2
Duration of Response (DOR) as assessed by local investigators | Up to 5 years
  Part 1 and Part 2
Odronextamab concentrations in serum when administered with CHOP | Up to 22 weeks
  Part 1 and Part 2
Occurrence of Anti-Drug Antibodies (ADA) to odronextamab | Up to 22 weeks
  Part 1 and Part 2
Magnitude of ADA to odronextamab | Up to 22 weeks
  Part 1 and Part 2
PFS assessed by local investigator review | Up to 5 years
  Part 2
EFS assessed by local investigator review | Up to 5 years
  Part 2
BOR assessed by ICR | Up to 22 weeks
  Part 2
DOR assessed by ICR | Up to 5 years
  Part 2
Incidence of TEAEs | Up to 2 years
  Part 2
Severity of TEAEs | Up to 2 years
  Part 2
Minimal Residual Disease (MRD) status | Up to 22 weeks
  Part 2
Change in physical functioning as measured by European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C) 30 | Up to 5 years
  Part 2 The EORTC QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional and social functioning), 3 symptom scales (fatigue, pain and nausea/vomiting), a GHS/QoL scale, and six single items (constipation, diarrhea, insomnia, shortness of breath, appetite loss and financial difficulties). For the functioning scales and global health status / QoL, scores range from 1 = "very poor" to 7 = "excellent" with higher scores indicate better functioning; for the symptom scales, scores range from 1 = "not at all" to 4 = "very much" higher scores indicate higher symptom burden.
Change in patient reported outcomes, as measured by EORTC QLQ-C30 | Up to 5 years
  Part 2 The EORTC QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional and social functioning), 3 symptom scales (fatigue, pain and nausea/vomiting), a GHS/QoL scale, and six single items (constipation, diarrhea, insomnia, shortness of breath, appetite loss and financial difficulties). For the functioning scales and global health status / QoL, scores range from 1 = "very poor" to 7 = "excellent" with higher scores indicate better functioning; for the symptom scales, scores range from 1 = "not at all" to 4 = "very much" higher scores indicate higher symptom burden.
Change in patient reported outcomes, as measured by Functional Assessment of Cancer Therapy - Lymphoma Subscale (FACT-LymS) | Up to 5 years
  Part 2 The FACT-Lym lymphoma subscale (LymS) includes 15 items to assess NHL-related symptoms and concerns. All questions are answered on a 5-point scale ranging from "not at all" (0) to "very much" (4). Higher scores are associated with a worse quality of life.
Change in patient reported outcomes, as measured by Patient Global Impression of Severity (PGIS) | Up to 5 years
  Part 2 The PGIS includes a single-item to assess how a patient perceives the overall severity of cancer symptoms over the past 7 days. Patients will choose the response that best describes the severity of their overall cancer symptoms with options on a 5-point scale ranging from 1 (No symptoms) to 4 (Very Severe).
Change in patient reported outcomes, as measured by Patient Global Impression of Change (PGIC) | Up to 5 years
  Part 2 The PGIC item includes a single-item to assess how a patient perceives their overall change in health status since the start of study treatment. Patients will choose from response options on a 7-point scale ranging from 1 (Much Better) to 7 (Much worse); 1- Much Better, 2-Moderately Better, 3-A Little Better, 4-About the Same, 5-A Little Worse, 6-Moderately Worse, 7-Much Worse.
Change in patient reported outcomes, as measured by EuroQol-5 Dimension-5 Level Scale (EQ-5D-5L) | Up to 5 years
  Part 2 The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: "no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems". The EQ VAS records the participant's self-rated health on a vertical visual analogue scale where the endpoints are labeled "Best imaginable health state" and "Worst imaginable health state".
Change in score of the Functional Assessment of Cancer Therapy-General (FACT-G ) GP5 item | Up to 5 years
  Part 2 A single item (GP5) of the validated FACT-G questionnaire will be used to assess from the participant perspective the overall impact of treatment side-effect. The question item is on a 5-point scale ranging from "not at all" (0) to "very much" (4).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (149):
- United States (18):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - University of California (UC) Davis, Sacramento, California
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - St Vincent Ascension at Peyton Manning Childrens Hospital, Indianapolis, Indiana
  - Investigative Clinical Research of Indiana, Noblesville, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Stony Brook University Hospital, Stony Brook, New York
  - Clinical Research Alliance Inc, Westbury, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Center for Oncology and Blood Disorders, Houston, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Prohealth Care Inc, Waukesha, Wisconsin
- Australia (5):
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Icon Cancer Centre - Wesley, Auchenflower, Queensland
  - Pindara Private Hospital, Benowa, Queensland
  - Epworth Freemasons, East Melbourne, Victoria
- Austria (6):
  - Landeskrankenhaus Hochsteiermark, Leoben, Styria
  - Kepler University Hospital, Linz, Upper Austria
  - Medical University Graz, Graz
  - Medical University of Vienna, Vienna
  - Hanusch Krankenhaus, Vienna
  - Klinikum Wels-Grieskirchen, Wels
- Belgium (5):
  - AZ St.-Elisabeth Herentals vzw, Herentals, Antwerp
  - Centre Hospitalier Regional de Verviers, Verviers, Liege
  - Universitair Ziekenhuis (UZ) Gent/ Ghent University Hospital, Ghent, Oost-Vlaanderen
  - Az Delta, Roeselare, West-Vlaanderen
  - Institut Jules Bordet, Brussels
- Chile (4):
  - Hospital Clinico Universidad de Los Andes, Santiago, Las Condes
  - Centro Oncologia de Precision Universidad Mayor, Santiago, Santiago Metropolitan
  - Inmunocel, Santiago, Santiago Metropolitan
  - Clinica Alemana de Santiago, Santiago
- Czechia (3):
  - University Hospital Hradec Kralove, Hradec Králové, East Bohemia
  - University Hospital Kralovske Vinohrady, Prague
  - Vseobecna Fakultni Nemocnice V Praze, Prague
- France (16):
  - Centre Hospitalier Universitaire (CHU) Rennes, Rennes, Brittany Region
  - CHRU de Tours, Tours, Centre-Val de Loire
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux, Gironde
  - Hopital Saint Vincent-de-Paul, Lille, Nord
  - Centre Hospitalier Universitaire (CHU) de Bordeaux, Pessac, Nouvelle-Aquitaine
  - Centre Hospitalier Universitaire De Poitiers, Poitiers, Nouvelle-Aquitaine
  - Nantes University Hospital, Nantes, Pays de la Loire Region
  - Centre Hospitalier Metropole Savoie, Chambéry, Savoie
  - Centre Hospitalier Universitaire Angers, Angers
  - Change Annecy, Metz-Tessy
  - CHU Nimes Institut de Cancerologie, Nîmes
  - Assistance Publique-Hopitaux de Paris (AP-HP), Paris
  - CHU de Saint-Etienne, Saint-Etienne
  - Hopital Victor Dupouy Argenteuil, Argenteuil, Île-de-France Region
  - Avicenne Hospital, Bobigny, Île-de-France Region
  - Gustave Roussy, Villejuif, Île-de-France Region
- Germany (8):
  - Robert-Bosch-Krankenhaus, Stuttgart, Baden-Wurttemberg
  - Kliniken Ostalb Stauferklinikum Schwab Gmund, Mutlangen, Gmund
  - Clinic Frankfurt (Oder), Frankfurt am Main, Hesse
  - University Hospital Essen, Essen, North Rhine-Westphalia
  - Universitaetsmedizin der Johannes Gutenberg Universitaet Mainz KoeR, Mainz, Rhineland-Palatinate
  - Hematological Praxis Dresden, Dresden, Saxony
  - University Hospital Carl Gustav Carus, Dresden
  - Stadtisches Krankenhaus Kiel, Kiel
- St James Hospital and Trinity College Dublin, Dublin, Ireland
- Israel (6):
  - The Chaim Sheba Medical Center, Tel Litwinsky, Tel Aviv
  - Samson Assuta Ashdod University Hospital, Ashdod
  - Bnai Zion Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (11):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Forli-Cesena
  - ASST Monza Ospedale San Gerardo, Monza, Monza E Brianza
  - Istituto Europeo di Oncologia, Milan
  - A.O.U. di Modena, Modena
  - Federico II University, Napoli
  - AOU Maggiore della Carita, Novara
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera di Perugia, Perugia
  - Ospedale Santa Maria delle Croci, Ravenna
  - Hematology - Città della Salute e della Scienza di Torino, Turin
  - Santa Maria della Misericordia, Udine
- Malaysia (5):
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Tg Ampuan Afzan, Kuantan, Pahang
  - Hospital Queen Elizabeth, Kota Kinabalu, Sabah
  - Hospital Ampang, Ampang, Selangor
  - Subang Jaya Medical Center, Subang Jaya, Selangor
- Poland (7):
  - Matopolskie Centrum Medyczne S.C., Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny, Wroclaw, Lower Silesian Voivodeship
  - Aidport, Skorzewo, Wielkopolska
  - Uniwersyteckie Centrum Kliniczne, Building of the Non-Invasive Medicine Center, Gdansk
  - Centrum Innowacyjnych Terapii Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Szpital Szpecjalistyczny w Walbrzychu, Wałbrzych
  - Wielospecjalistyczne Centrum Onkologii i Traumatologii, Lodz, Łódź Voivodeship
- Singapore (3):
  - National University Hospital Singapore, Singapore
  - National Cancer Centre of Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (11):
  - St. Vincent Hospital - The Catholic University of Korea, Suwon, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Namdong-Gu
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Yeyungnam University Medical Center, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Yeouido St. Marys Hospital, Seoul
  - Seoul St Marys Hospital, Seoul
- Spain (19):
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Son Espases University Hospital, Palma, Balearic Islands
  - Hospital Universitari Parc Tauli, Sabadell, Barcelona
  - Hospital Universitari Mutua Terrassa, Terrassa, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Sant Pau, Barcelona
  - Hospital Virgen De Las Nieves De Granada, Granada
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Fundacion Jimenez Diaz University Hospital, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Instituto Valenciano de Oncologia, Valencia
  - University Hospital Doctor Peset, Valencia
  - Universitat de Valencia - Hospital Universitari i Politecnic La Fe de Valencia (Hospital La Fe Bulevar Sur), Valencia
- Taiwan (6):
  - Chang Gung Medical Foundation Chia Yi Branch, Buzi, Chiayi County
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan District, Hunan Province
  - Changhua Christian Hospital, Changhua
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - Wanfang Hospital, Taipei
  - National Taiwan University Hospital, Taipei
- Thailand (4):
  - Chulalongkorn University, Bangkok, Krung Thep Maha Nakhon [Bangko]
  - Sriraj Hospital, Bangkok
  - Chaing Mai University, Chiang Mai
  - Faculty of Medicine, Khon Kaen
- Turkey (Türkiye) (9):
  - Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Yenimahalle, Ankara
  - VM Medical Park Mersin Hospital, Mezitli, Mersin
  - Tekirdag Namik Kemal University Hospital, Tekirdağ, Suleymanpasa
  - Gazi Universitesi, Beşevler
  - Istanbul University Istanbul Faculty of Medicine, Istanbul
  - Ege University, Izmir
  - Dokuz Eylul University, Izmir
  - Sakarya University Medical Faculty, Sakarya
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
- United Kingdom (2):
  - NHS Grampian: Aberdeen Royal Infirmary, Aberdeen
  - The Hillingdon Hospitals NHS Foundation Trust, Uxbridge

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: OLYMPIA — https://olympiastudies.com/en-us